CLINICAL TRIAL: NCT07336862
Title: The Efficacy and Safety of Bariatric Surgery Combined With GLP-1 Receptor Agonists for Patients With Severe Obesity: A Prospective, Multicenter Cohort Study
Brief Title: Bariatric Surgery Combined With GLP-1 Receptor Agonists Study
Acronym: BS-GLP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Prof., China-Japan Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-339
Record Dates: First submitted 2025-09-29; First posted 2026-01-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: obesity; Glucagon-Like Peptide-1 Receptor Agonists; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BS-GLP group (Experimental): Names for Surgery: Laparoscopic Sleeve Gastrectomy. Names for drugs: Semaglutide. Dosage:The starting dose was 0.25 mg per week and was subsequently titrated up based on individual patient response to a maximum maintenance dose of 2.4 mg per week.
  Frequency: Once per week. Duration: The treatment continued until the completion of the 6-month postoperative period.
  Interventions: Combination Product: BS-GLP group
- BS group (Other): Names for Surgery: Laparoscopic Sleeve Gastrectomy. Names for drugs: N/A. Observation Group: Received only basic nutritional recommendation interventions after surgery.
  Interventions: Procedure: BS group

INTERVENTIONS:
Combination Product: BS-GLP group — 1. Basic Treatment Measures Within 0-30 days after sleeve gastrectomy, all patients received very low-calorie enteral nutrition powder (100 kcal/day). From 30 to 90 days post-surgery, a low-energy diet (400 kcal/day) was provided. Beyond 90 days post-surgery, a calorie-restricted diet was implemented (1,500 kcal/day for men and 1,200 kcal/day for women).
  2. In addition to laparoscopic sleeve gastrectomy and postoperative basic nutritional counseling,the intervention group received subcutaneous semaglutide injections from 1 to 6 months postoperatively.The specific protocol was as follows:In the intervention group, semaglutide treatment was initiated at 1 month after LSG. The starting dose was 0.25 mg per week and was subsequently titrated up based on individual patient response to a maximum maintenance dose of 2.4 mg per week. The treatment continued until the completion of the 6-month postoperative period.
  Arms: BS-GLP group
Procedure: BS group — 1. Basic Treatment Measures Within 0-30 days after sleeve gastrectomy, all patients received very low-calorie enteral nutrition powder (100 kcal/day). From 30 to 90 days post-surgery, a low-energy diet (400 kcal/day) was provided. Beyond 90 days post-surgery, a calorie-restricted diet was implemented (1,500 kcal/day for men and 1,200 kcal/day for women).
  2. Observation Group: Received only basic nutritional recommendation interventions after surgery.
  Arms: BS group

SUMMARY:
Obese patients exhibit considerable heterogeneity and complex comorbidities, making long-term effective management challenging with single therapies. While bariatric surgery remains the most effective weight-loss intervention, postoperative weight regain and metabolic deterioration require attention. GLP-1 RAs offer distinct advantages for weight and metabolic improvement, and their combined application with surgery may yield synergistic benefits. This study investigates the efficacy and safety of bariatric surgery combined with GLP-1 receptor agonist adjuvant therapy for severe obesity.

DETAILED DESCRIPTION:
"bariatric surgery is guideline-recommended as an effective obesity treatment. Substantial evidence demonstrates its ability to significantly reduce weight, improve comorbidities like type 2 diabetes (T2DM) and dyslipidemia, and lower cardiovascular risk. However, the significant heterogeneity and complex comorbidity profiles among obese patients challenge long-term effective management with single therapeutic approaches. While currently the most effective weight-loss intervention, bariatric surgery requires attention to issues such as postoperative weight regain and metabolic deterioration.

In parallel, Glucagon-like peptide-1 receptor agonists (GLP-1RA) have demonstrated significant efficacy in obesity management. Agents like semaglutide promote weight loss and metabolic improvement through mechanisms including insulin secretion promotion, appetite suppression, delayed gastric emptying, and enhanced satiety.

Given the distinct advantages of both bariatric surgery and GLP-1RA therapy in weight and metabolic control, this study will combine these modalities into a comprehensive treatment strategy. The investigators will compare the long-term safety and effectiveness of different combination regimens for weight management and metabolic improvement in patients with severe obesity."

ELIGIBILITY:
Inclusion Criteria:

1. Primary metabolic surgery candidates: Patients undergoing initial laparoscopic sleeve gastrectomy (LSG)
2. obesity:BMI ≥35 kg/m²
3. Metabolic comorbidities: Diagnosis of metabolic syndrome or type 2 diabetes mellitus (T2DM) meeting standard criteria
4. Age range: 18-60 years (inclusive)
5. Informed consent: Willing participation with documented consent

Exclusion Criteria:

1. Recent GLP-1RA use: Treatment with GLP-1 receptor agonists within 6 months preoperatively
2. Prior bariatric surgery: History of any metabolic/bariatric surgical procedure
3. Postoperative complications: Requiring reoperation for severe complications (e.g., hemorrhage, anastomotic leak)
4. Non-indicated candidates: Patients not meeting standard bariatric surgery indications
5. Significant comorbidities:

   * Advanced hepatic/renal dysfunction (Child-Pugh C or eGFR <30 mL/min/1.73m²)
   * Active malignancy (except non-melanoma skin cancers)
   * Autoimmune disorders requiring immunosuppression
   * Uncontrolled psychiatric conditions (e.g., active psychosis, severe depression)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the Percentage of weight loss | 1 year
  Through study completion, an average of 1 year, the investigators will observe the Percentage of weight loss.

SECONDARY OUTCOMES:
body fat percentage(BFP) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Gender | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Ethnicity | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Height in meters | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Visceral fat area | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Weight in kilograms | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Waist circumference in centimeters | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Hip circumference in centimeters | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Blood pressure | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Muscle mass in kilograms | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Body fat percentage | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Serum creatinine | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Glomerular filtration rate | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Fasting blood glucose | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Average blood glucose from continuous glucose monitoring | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Postprandial 2-hour blood glucose | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
HbA1c | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Urinary microalbumin and other Urinalysis indexes | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Total cholesterol | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Low-Density Lipoprotein(LDL) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
High-Density Lipoprotein(HDL) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Triglycerides | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Alanine Aminotransferase(ALT) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
Aspartate Aminotransferase(AST) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
lean body mass (LBM) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
lean body mass percentage (LBMP) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
urine microalbumin-to-creatinine ratio (ACR) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.
uric acid(UA) | Immediately postoperatively (Day 0), and at 1, 3, 6, and 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Meng, Ph.D, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China